CLINICAL TRIAL: NCT05227183
Title: Prevention of Suicidal Behavior Through the VIGILANS Protocol: the Restoration of Social Connection Hypothesis
Acronym: RECONEX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RECMPL21_0405
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Suicidal Behaviour Disorder
Keywords: suicide; social stress; suicide monitoring; cardiovascular; neuroendocrinology
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Masking Description: non applicable
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with suicidal recurrence during VigilanS monitoring (Reattempters) (Experimental): Patients with at least a past experience of suicidal attempt (SA), included after their last SA in the 6 months VigilanS monitoring protocol and who have presented a recurrence of SA during this monitoring
  Interventions: Behavioral: The virtual version of the Social stress task : V-TSST
- Patients without suicidal recurrence during VigilanS monitoring (No reattempters) (Experimental): Patients with at least a past experience of suicidal attempt (SA), included after their last SA in the 6 months VigilanS monitoring protocol and who have not presented a recurrence of SA during this monitoring
  Interventions: Behavioral: The virtual version of the Social stress task : V-TSST

INTERVENTIONS:
Behavioral: The virtual version of the Social stress task : V-TSST — The task consists in a brief presentation about the abilities of participants followed by an arithmetic task in front of a virtual 3D audience projected and one researcher in a room.First, participants have 5 minutes to prepare an exhibition about their qualities, their strengths and defects, and, why they identify with them. During this period virtual reality shows a closed curtain, and sounds from the audience can be heard. In the second phase, the curtain is raised and the participant must expose his speech during 5 minutes. Audience will remain attentive during 2 minutes, then audience will change to a restless attitude. The third phase consists of subtracting back a two-digit number from a four-digit number, as quickly as possible, starting again if participant makes a mistake. A debriefing of the test is scheduled at the end of the protocol, to remind patients of the purely fictional nature of this test. The visit will only end after a return to the baseline emotional state

SUMMARY:
The World Health Organization (WHO) estimates, with 800,000 annual deaths, that suicide is the second leading cause of death in people aged 10 to 44 and thus recognizes suicide prevention as a public health priority. The psychological impact of the COVID-19 pandemic, the social isolation and the economic consequences engendered by the confinement, as well as the direct effects of this viral infection increase suicidal mortality.

Sensitivity to social rejection in suicide : Epidemiological and clinical studies indicate that social isolation and loneliness are very strongly associated with suicide. Our works suggests that suicide vulnerability is associated with specific processing of social information related to brain regions playing a role in psychological pain and inflammation. In fact, social stresses are powerful inducers of inflammation, also associated with suicide. Thus, we hypothesize that patients at risk of suicide could be particularly sensitive to social adversity (social stress / lack of social support), via the activation of specific brain regions regulating social cognitions, psychological pain and 'inflammation.

The VigilanS device: a monitoring tool in suicide prevention. VigilanS is a national telephone recontact system initiated in 2015, which has already shown its effectiveness in preventing suicidal recurrence. Patients admitted to the Emergency Department of the Montpellier and Nimes CHUs for SA benefit from VigilanS monitoring for 6 months (period of major risk). These organized calls aim to assess the patient's condition, manage a possible suicidal crisis and ensure the compromise for discharge from the emergency room. It is important to determine the factors explaining the effectiveness of this device.

Thus, we formulate the hypothesis that VigilanS prevents suicidal recurrence by acting on the restoration of the social bond in subjects vulnerable to suicide and isolated. We will test the hypothesis that the preventive effect of the VigilanS device on suicidal recurrence during the 6 months of the day before depends on the sensitivity to social stress of the suicidal patients (measured by the response to an experimental task of social stress).

DETAILED DESCRIPTION:
Main Objective :

To compare the cortisol response to an experimental social stress task, the virtual trier social stress test (V-TSST), between patients who performed a relapse in suicide attempt (TS+) vs. did not relapsed (TS-) during the VigilanS monitoring .

Secondary Objectives :

1. To compare the biological (alpha amylase and inflammatory markers), cardiac (heart rate variability), and emotional response to an experimental social stress task (V-TSST), between patients who reattempted suicide (TS+) vs. those that did not (TS-) during the VigilanS monitoring;
2. Demonstrate that social support, feelings of loneliness and isolation are associated with the prevention of suicidal relapse during VigilanS;
3. Demonstrate that social cognition performance is associated with the prevention of suicidal recidivism during VigilanS;
4. To assess the predictive value of the experimental social stress response regarding suicidal relapse during an additional 6 months of follow-up (without VigilanS monitoring)

It is an interventional research, multicentric, which involves only minimal risks and constraints.

We will recruit 120 patients who had performed a suicide attempt according to the Columbia-suicide severity rating scale (C-SSRS) and were included in VigilanS.

* 60 patients who had a suicidal recurrence during the 6 months of the VigilanS monitoring protocol (TS+) according to the Columbia-suicide severity rating scale (C-SSRS).
* 60 patients who had not suffered a suicidal recurrence during the 6 months of the VigilanS monitoring protocol (TS-).

Patient participation includes 3 visits : inclusion visit (clinical ans psychological assessment), experimental Visit (V-TSST with cardiovascular, neuroendocrine, inflammatory measures), 6months follow up visit to assess suicidal recurrence

Perspectives : This study will contribute to a better understanding of the pathophysiological mechanisms of suicidal behavior in a social stress environment. The results could help us to prevent suicidal behavior in the most vulnerable individuals and, potentially, to develop a therapeutic approach complementary to VigilanS such as biofeedback and mindfulness interventions in difficult situations so that patients can better adapt to social stressors in real life.

ELIGIBILITY:
For all subjects:

* Patients benefiting from VigilanS monitoring at CHU Montpellier / Nîmes
* aged between 18 and 55 years old;
* able to understand experimental procedures
* able to speak, read and understand French
* able to give written informed consent

Specific inclusion criteria:

TS+: Had an actual suicide according to C-SSRS suicidal recurrence during the 6 months prior to VigilanS

TS-: Had not suffered a suicidal recurrence during the 6 months prior to VigilanS

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2027-03-13 (Estimated); Study Completion 2027-09-13 (Estimated)

PRIMARY OUTCOMES:
Change in salivary cortisol | Visit 2 : between 0 to 7 days after inclusion
  study of the change in salivary cortisol, across all procedure (from -10 to +15, +30, +45 and +60 minutes following the completion of V-TSST)

SECONDARY OUTCOMES:
Changes in cardiovascular response (heart rate) | Visit 2 : between 0 to 7 days after inclusion
  study of the changes in heart rate (HR) from -10 to +15, +30, +45 and +60 minutes following the completion of V-TSST.
Changes in cardiovascular response (Cardiac output) | Visit 2 : between 0 to 7 days after inclusion
  study of the changes in Cardiac output (CO) from -10 to +15, +30, +45 and +60 minutes following the completion of V-TSST.
Changes in cardiovascular response (Total peripheral resistance) | Visit 2 : between 0 to 7 days after inclusion
  study of the changes in Total peripheral resistance (TPR) from -10 to +15, +30, +45 and +60 minutes following the completion of V-TSST.
Changes in cardiovascular response (time between the two R peaks) | Visit 2 : between 0 to 7 days after inclusion
  study of the changes in time between the two R peaks(time between the two R peaks) from -10 to +15, +30, +45 and +60 minutes following the completion of V-TSST.
Changes in cardiovascular response (pre-ejection period) | Visit 2 : between 0 to 7 days after inclusion
  study of the changes in pre-ejection period (PEP) from -10 to +15, +30, +45 and +60 minutes following the completion of V-TSST.
Changes in cardiovascular response (Vascular contractibility) | Visit 2 : between 0 to 7 days after inclusion
  study of the changes in vascular contractibility (VC) from -10 to +15, +30, +45 and +60 minutes following the completion of V-TSST.
Changes in cardiovascular response (High frequency) | Visit 2 : between 0 to 7 days after inclusion
  study of the changes in High frequency (HF) from -10 to +15, +30, +45 and +60 minutes following the completion of V-TSST.
Changes in cardiovascular response (Low frequency) | Visit 2 : between 0 to 7 days after inclusion
  study of the changes in Low frequency (LF) from -10 to +15, +30, +45 and +60 minutes following the completion of V-TSST.
Changes in cardiovascular response (Very low frequency) | Visit 2 : between 0 to 7 days after inclusion
  study of the changes in Very low frequency (VLF) from -10 to +15, +30, +45 and +60 minutes following the completion of V-TSST.
Changes in cardiovascular response (Root mean squared of successive R-R interval differences) | Visit 2 : between 0 to 7 days after inclusion
  study of the changes in Root mean squared of successive R-R interval differences (RMSSD) from -10 to +15, +30, +45 and +60 minutes following the completion of V-TSST.
Changes in salivary α-amylase | Visit 2 : between 0 to 7 days after inclusion
  Study of the changes in salivary α-amylase, after V-TSST, from -10 to +15, +30, +45 and +60 minutes following the completion fo V-TSST
Risk Taking decision making after V-TSST | Visit 2 : between 0 to 7 days after inclusion
  risk-taking using Iowa Gambling (IG) index from Iowa Gambling Task (IGT)
Sense of fairness/unfairness after V-TSST | Visit 2 : between 0 to 7 days after inclusion
  Using the total score of Ultimatum
Prissoner's Dilemma | Visit 2 : between 0 to 7 days after inclusion
  Using the sum of A choice´s
Reading the mind in the eyes | Visit 2 : between 0 to 7 days after inclusion
  Using the percentage of correct answer in the test
Changes in anxiety level induced by V-TSST | Visit 2 : between 0 to 7 days after inclusion
  Changes in psychometric state measures : anxiety using the state anxiety inventory, after V-TSST, from -10 to + 15, + 60 and + 120 minutes post V-TSST
Changes in depression level induced by V-TSST | Visit 2 : between 0 to 7 days after inclusion
  Changes in psychometric state measures : mood using the Positive and Negative Affect Schedule, after V-TSST, from baseline to + 15, + 60 and + 120 minutes post V-TSST
Changes in psychological pain level induced by V-TSST | Visit 2 : between 0 to 7 days after inclusion
  Changes in psychometric state measures : psychological pain using a visual analogue scale, after V-TSST, from baseline to + 15, + 60 and + 120 post V-TSST. The score ranges from 0 to 10, a higher score indicates the most important psychological pain
Changes in suicidal ideation level induced by V-TSST | Visit 2 : between 0 to 7 days after inclusion
  Changes in psychometric state measures : suicidal ideation using a visual analogue scale, after V-TSST, from baseline to + 15, + 60 and + 120 post V-TSST. SST. The score ranges from 0 to 10, a higher score indicates the most important suicidal ideation
Changes in social distress level induced by V-TSST | Visit 2 : between 0 to 7 days after inclusion
  Changes in psychometric state measures : social distress using a visual analogue scale, after V-TSST, from -10 to + 15, + 60 and + 120 minutes post V-TSST. The score ranges from 0 to 10, a higher score indicates the most important social distress
Changes in C-Reactive Protein (CRP) induced by V-TSST | Visit 2 : between 0 to 7 days after inclusion
  Study of the changes in CRP, after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in Interleukin (IL) - 1b induced by V-TSST | Visit 2 : between 0 to 7 days after inclusion
  Study of the changes in Interleukin (IL) - 1b after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in IL-6 induced by V-TSST | Visit 2 : between 0 to 7 days after inclusion
  Study of the changes in IL-6 after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in IL1β induced by V-TSST | Visit 2 : between 0 to 7 days after inclusion
  Study of the changes in IL1β after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in IL4 induced by V-TSST | Visit 2 : between 0 to 7 days after inclusion
  Study of the changes in IL4 after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in IL8 induced by V-TSST | Visit 2 : between 0 to 7 days after inclusion
  Study of the changes in IL8 after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in IL10 induced by V-TSST | Visit 2 : between 0 to 7 days after inclusion
  Study of the changes in IL10 after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in IL13 induced by V-TSST | Visit 2 : between 0 to 7 days after inclusion
  Study of the changes in IL13 after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in IL27 induced by V-TSST | Visit 2 : between 0 to 7 days after inclusion
  Study of the changes in IL27 after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in NF-KB protein induced by V-TSST | Visit 2 : between 0 to 7 days after inclusion
  Study of the changes in NF-KB protein after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in IKB protein induced by V-TSST | Visit 2 : between 0 to 7 days after inclusion
  Study of the changes in IKB protein after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in Tumor necrosis factor (TNF) - α protein induced by V-TSST | Visit 2 : between 0 to 7 days after inclusion
  Study of the changes in Tumor necrosis factor (TNF) - α protein after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in Interferon (IFN) - γ induced by V-TSST | Visit 2 : between 0 to 7 days after inclusion
  Study of the changes in Interferon (IFN) - γ after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in Vascular endothelial growth factor (VEGF) induced by V-TSST | Visit 2 : between 0 to 7 days after inclusion
  Study of the changes in Vascular endothelial growth factor (VEGF) after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in kyrunenine induced by V-TSST | Visit 2 : between 0 to 7 days after inclusion
  Study of the changes in kyrunenine after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in sCD62P induced by V-TSST | Visit 2 : between 0 to 7 days after inclusion
  Study of the changes in sCD62P after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in sCD40L induced by V-TSST | Visit 2 : between 0 to 7 days after inclusion
  Study of the changes in sCD40L after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in Platelet factor (PF) 4 induced by V-TSST | Visit 2 : between 0 to 7 days after inclusion
  Study of the changes in PF4 after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in RANTES induced by V-TSST | Visit 2 : between 0 to 7 days after inclusion
  Study of the changes in RANTES after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in Brain derived neurotrophic factor (BDNF) induced by V-TSST | Visit 2 : between 0 to 7 days after inclusion
  Study of the changes in BDNF after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in sOx40L induced by V-TSST | Visit 2 : between 0 to 7 days after inclusion
  Study of the changes in sOx40L after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in Microparticle induced by V-TSST | Visit 2 : between 0 to 7 days after inclusion
  Study of the changes in Microparticle after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
Changes in Mitochondrial DNA of platelet origin induced by V-TSST | Visit 2 : between 0 to 7 days after inclusion
  Study of the changes in Mitochondrial deoxyribonucleic acid (DNA) of platelet origin after the V-TSST, from -10 to +15, +60, +90 and +120 minutes following the completion post V-TSST.
loneliness levels | inclusion Visit
  Study of response to V-TSST depending on basal loneliness levels assed by UCLA Loneliness Scale. A higher score indicates high loneliness levels
Perceived social support | inclusion Visit
  Study of response to V-TSST depending on basal perceived social support levels assed by the "Questionnaire de Soutien Social Perçu" . A higher score indicates high perception of social support
Availability of social support | inclusion Visit
  Study of response to V-TSST depending on basal levels of social support assed by the Social Provisions Scale . A higher score indicates high availability of social support
Perceived online social support | inclusion Visit
  Study of response to V-TSST depending on basal levels of online social support assed by the online social support scale . A higher score indicates high perception of online social support
Social isolation | inclusion Visit
  Study of response to V-TSST depending on basal levels of social isolation assed by the Steptoe Social Isolation scale . A higher score indicates high perception of online social support
Suicidal recurrence | 6months follow up Visit
  Occurrence of a suicidal event within 6 months of study follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Maude SENEQUE, Montpellier, France